CLINICAL TRIAL: NCT04705389
Title: SerUM Markers in MERkel Cell Carcinoma Patients: a Longitudinal moniTorIng Study for optiMization of European Guidelines
Acronym: SUMMERTIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: European Academy of Dermatology and Venerology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DR200079
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2020-11

CONDITIONS: Merkel Cell Carcinoma
Keywords: biomarker; monitoring; prognosis; merkel cell polyomavirus; miR375; T-antigen antibodies
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case group (Other): Intervention only includes additional blood sampling at baseline and during follow up (5 samplings).
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — blood samples

SUMMARY:
Merkel cell carcinoma (MCC) is a rare aggressive skin carcinoma. Approximately 80% of MCC are related to the Merkel Cell Polyomavirus (MCPyV). Although rates of relapse are high, the follow-up strategy lacks consensus. Patients are usually assessed clinically every 3 to 6 months for the first 2-3 years, and every 6 to 12 months thereafter. In the European guidelines, patients with early stages are monitored with clinical examination and ultrasonography of lymph nodes, while whole-body imaging is optional in patients with stage III disease, on a yearly basis for 5 years. Such strategy may prevent the diagnosis of infra-clinical recurrences, whereas patients could still be treated with surgery or radiation therapy. Until 2017, patients with advanced disease were treated with chemotherapies, with no long-term benefit. Immunotherapies with PD-1/PD-L1 inhibitors currently allow durable responses in 50% of such patients. This major change in the management of MCC patients argues for a follow-up strategy that would allow early diagnosis of infra-clinical metastases, when tumoral burden is still low. Given that all patients cannot be monitored by systematic regular imaging, additional non-invasive tools are needed. Blood-based biomarkers as a surrogate of tumor burden are advantageous as they can be repeated over time, providing guidance on when imaging is necessary. The study aims to assess two blood biomarkers, MCPyV T-Ag antibodies and cell-free miR-375, in a prospective fashion from baseline diagnosis, in a cohort of 150 European MCC patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with a " de novo " diagnosis of MCC, confirmed on histological criteria (neuroendocrine morphology, CK20 staining and/or neuroendocrine and/or SATB2 staining, exclusion of differential diagnosis)
* ≥ 18 years of age
* Written informed consent obtained from the participant

Exclusion Criteria:

* Patients following any measures of legal presentation
* Pregnancy or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
To assess the diagnostic performances of two blood biomarkers (T-antigen antibodies and miR375) in detecting disease recurrence during follow up of patients with Merkel Cell Carcinoma | 12 months
  Diagnostic performances (specificity, sensitivity, predictive values) of each biomarker will be assessed at the end of follow up, in relation with patients' outcomes (remission and recurrence).

SECONDARY OUTCOMES:
To assess if these two blood biomarkers (T-antigen antibodies and miR375) assessed at baseline are associated with prognosis and response to treatments. | 12 months
  Cox regression analysis will be performed to evaluate the clinical and biological factors associated with recurrence, death of disease, response to treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Mahtab SAMIMI, MD-PhD, Study Director — University Hospital, Tours
Locations (10):
- Department of Dermatology, Medical University of Vienna, Vienna, Austria
- University Hospital of Helsinki, Finland, Helsinki, Finland
- Dermatology Dept, Hospital University of Tours, Tours, France
- Translational Skin Cancer Research, Essen, Germany
- National Tumour Institute "Fondazione G. Pascale" Unit of Melanoma - Cancer Immunotherapy and Innovative therapy, Naples, Italy
- Academic Hospital of Maastricht, Maastricht, Netherlands
- Department of Dermatology, Carol Davila University of Medicine and Pharmacy, Bucharest, Romania
- Skin Cancer and Surgery Center, Sahlgrenska University Hospital, Gothenburg, Sweden
- Department of Dermatology, Başkent University Faculty of Medicine, Ankara, Turkey (Türkiye)
- Queen Elizabeth Hospital, Birmingham, United Kingdom

REFERENCES:
- [Background] Fan K, Ritter C, Nghiem P, Blom A, Verhaegen ME, Dlugosz A, Odum N, Woetmann A, Tothill RW, Hicks RJ, Sand M, Schrama D, Schadendorf D, Ugurel S, Becker JC. Circulating Cell-Free miR-375 as Surrogate Marker of Tumor Burden in Merkel Cell Carcinoma. Clin Cancer Res. 2018 Dec 1;24(23):5873-5882. doi: 10.1158/1078-0432.CCR-18-1184. Epub 2018 Jul 30. PMID 30061360
- [Background] Kervarrec T, Tallet A, Miquelestorena-Standley E, Houben R, Schrama D, Gambichler T, Berthon P, Le Corre Y, Hainaut-Wierzbicka E, Aubin F, Bens G, Tabareau-Delalande F, Beneton N, Fromont G, Arbion F, Leteurtre E, Touze A, Samimi M, Guyetant S. Diagnostic accuracy of a panel of immunohistochemical and molecular markers to distinguish Merkel cell carcinoma from other neuroendocrine carcinomas. Mod Pathol. 2019 Apr;32(4):499-510. doi: 10.1038/s41379-018-0155-y. Epub 2018 Oct 22. PMID 30349028
- [Background] Paulson KG, Lewis CW, Redman MW, Simonson WT, Lisberg A, Ritter D, Morishima C, Hutchinson K, Mudgistratova L, Blom A, Iyer J, Moshiri AS, Tarabadkar ES, Carter JJ, Bhatia S, Kawasumi M, Galloway DA, Wener MH, Nghiem P. Viral oncoprotein antibodies as a marker for recurrence of Merkel cell carcinoma: A prospective validation study. Cancer. 2017 Apr 15;123(8):1464-1474. doi: 10.1002/cncr.30475. Epub 2016 Dec 7. PMID 27925665
- [Background] Samimi M, Molet L, Fleury M, Laude H, Carlotti A, Gardair C, Baudin M, Gouguet L, Maubec E, Avenel-Audran M, Esteve E, Wierzbicka-Hainaut E, Beneton N, Aubin F, Rozenberg F, Dupin N, Avril MF, Lorette G, Guyetant S, Coursaget P, Touze A. Prognostic value of antibodies to Merkel cell polyomavirus T antigens and VP1 protein in patients with Merkel cell carcinoma. Br J Dermatol. 2016 Apr;174(4):813-22. doi: 10.1111/bjd.14313. Epub 2016 Feb 3. PMID 26600395